CLINICAL TRIAL: NCT05736887
Title: Exploratory Efficacy of N-Acetylcysteine in Patients With History of COVID-19
Acronym: NACoV
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, RICHELDI LUCA, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 499
Record Dates: First submitted 2023-02-20; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-Acetylcysteine arm (Experimental): Subjects with recent history of COVID-19 infection randomized to receive N-Acetylcysteine.
  Interventions: Drug: N-Acetylcysteine
- Placebo arm (Placebo Comparator): Subjects with recent history of COVID-19 infection randomized to receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-Acetylcysteine — N-Acetylcysteine in 600mg tablets
  Arms: N-Acetylcysteine arm
Drug: Placebo — Placebo in 600mg tablets
  Arms: Placebo arm

SUMMARY:
A randomized, double-blind, parallel-arm, phase II, explorative study investigating the efficacy and safety of orally administered N-Acetylcysteine (NAC) versus placebo in patients with history of SARS-Cov-2 infection and residual respiratory impairment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤90 years.
2. History of hospitalization for COVID-19 pneumonia, as documented by positive RT/PCR testing for SARS-Cov-2 infection (nasopharyngeal swab) and suggestive radiological findings at the chest CT scan.
3. Resolution of SARS-CoV-2 infection as defined by negative RT/PCR testing (nasopharyngeal swab).
4. Evidence of residual interstitial lung abnormalities (including any of the following: ground glass, reticulation, or consolidation with overall extent ≥5% of total lung volume) on chest high resolution CT scan (performed during screening or within 30 days from screening visit) AND

One or more of the following:

* DLco ≤ 70 % of predicted value at screening
* Oxygen desaturation at 6-minute walk test (6MWT) ≥4% from baseline value at screening.
* Total Lung Capacity ≤ 80 % of predicted value at spirometry performed at screening
* Exertional dyspnea at screening, as defined by MMRC ≥1

Exclusion Criteria:

1. Evidence of resting respiratory failure, as defined by PaO2 ≤60 mmHg (FiO2 21%) at blood gas analysis at screening.
2. History of interstitial lung disease, or evidence of interstitial lung disease at screening that suggests any of the following: idiopathic interstitial pneumonias; lung diseases related to exposure to fibrogenic agents or other environmental toxins or drugs; other types of occupational lung diseases; granulomatous lung diseases; pulmonary vascular diseases; systemic diseases, including vasculitis, infectious diseases (Other than SARS-Cov-2 infection) and connective tissue diseases.
3. History of other types of respiratory diseases, including disorders of the airways, lung parenchyma, pleural space, mediastinum, diaphragm, or chest wall that, in the opinion of the Investigator, would impact the primary protocol endpoint or otherwise preclude the subject's participation in the study.
4. Any other known disease, medical conditions or blood test abnormalities that in the opinion of the Investigator may put the patient at risk because of participation, interfere with study procedures or cause concern regarding the patient inability to participate in the study.
5. Concomitant treatment with oral corticosteroids and/or other immunosuppressive drugs.
6. Pregnancy status.
7. Incapacity of providing valid informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
DLco | Week 12
  Change in percent predicted DLco at week 12 compared to baseline

SECONDARY OUTCOMES:
DLco | Week 12
  Change in absolute (ml/min/mmHg) predicted DLco from baseline to week 12
St. George's Respiratory Questionnaire (SGRQ) | Week 12
  Change in St. George's Respiratory Questionnaire (SGRQ) score from baseline to week 12.
Shortness of Breath Questionnaire (UCSD-SOBQ) | Week 12
  Change in University of California San Diego - Shortness of Breath Questionnaire (UCSD-SOBQ) score from baseline to week 12.
Change in Leicester Cough Questionnaire (LCQ) | Week 12
  Change in Leicester Cough Questionnaire (LCQ) from baseline to week 12.
Forced Vital Capacity (FVC) | Week 12
  Change in FVC (L) from baseline to week 12.
High-resolution computed tomography (HRCT) | Week 12
  Proportion of patients with improvement of interstitial changes on chest high-resolution computed tomography at 12 weeks, as defined by central radiological review.
Quantitative Lung Fibrosis | Week 12
  Change in Quantitative Lung Fibrosis (QLF) volume from baseline to week 12.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Agostino Gemelli IRCCS, Rome, Roma, Italy

IPD SHARING:
Plan to Share IPD: No